CLINICAL TRIAL: NCT01090284
Title: The Immunologic Reaction to Polypropylene Mesh Implantation: a Comparison Between Heavyweight and Lightweight Mesh.
Brief Title: The Immunologic Reaction to Polypropylene Mesh in Inguinal Hernioplasty
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Catania (Other)
Responsible Party: Prof. Angelo Donati, University of Catania
Other Study IDs: CH001GENI
Record Dates: First submitted 2010-03-18; First posted 2010-03-19 (Estimated); Last update posted 2010-03-23 (Estimated); Status verified 2010-02

CONDITIONS: Inguinal Hernia
Keywords: Inguinal hernia; Immune system; Cytokines; Prosthetic repair; Oxidative Stress
MeSH Terms: conditions — Hernia, Inguinal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Heavy weight mesh: This cohort includes patients undergoing inguinal hernioplasty with polypropylene heavy weight mesh.
  Interventions: Device: Inguinal hernioplasty
- Light weight mesh: This cohort includes patients undergoing inguinal hernioplasty with polypropylene light weight mesh.
  Interventions: Device: Inguinal hernioplasty

INTERVENTIONS:
Device: Inguinal hernioplasty — A conventional Prosthetic Inguinal Hernioplasty (Trabucco's Technique) will be performed by using polypropylene mesh.

SUMMARY:
The notable development and diffusion of prosthetic surgery of the abdominal wall over the last few years has led to the introduction of light weight meshes. The efficacy of inguinal hernia repair with light weight prosthesis, as well as the better or worse biotolerability with respect to those of light weight, remains questionable in literature, where a clear answer still remains to be given. If there exists a connection between the quantity of material implanted, the immunological reaction to the mesh, the induced oxidative stress and the degree of cicatrization, and consequently the long-term result of the efficacy of the operation, remains to be demonstrated. There are few studies on the immunological reaction to polypropylene meshes, and none on the oxidative stress induced by the mesh. Moreover, only one study has been published that clearly correlates the immunological reaction to the amount of prosthetic material, but was carried out on only a few patients.

The aim of this research is to show if there is a relationship between the amount of prosthetic material used and immunological reactions as well as postoperative oxidative stress, and thus to evaluate, if present, the differences in the biological reaction and biotolerability between light-weight and heavy-weight meshes on a statistically significant number of patients.

DETAILED DESCRIPTION:
Double blind randomization. The recruitment of patients will take place in the order that they are referred to the hernia service of the General Surgery and Week Surgery Unit of the University Hospital of Catania. After the examination confirming the diagnosis of inguinal hernia and once surgery has be indicated, informed consent will be obtained from the patient by means of a standardized form. The assignment to group H or group L will be made following a simple criterion of alternation that is completely random: i.e. patient 1 (Group H), patient 2 (Group L).A total of 60 patients will be recruited and divided into the two groups. For group H inguinal hernioplastic surgery will be carried out with the so called "heavy-weight" mesh (about 220 g/m2 of polypropylene), for Group L, on the other hand, the mesh will be of the "light-weight" type (about 40 g/m2).

A preoperative blood test will be carried out to determine the basal levels of IL-6, TNF-alpha, nitrites, GSH and isoprostanes) and 3 postoperative tests (at 6 h, 3 days and 12 days), all samples will be frozen for reference.

All the data from each patient will be collected in a personal file compiled by the surgeon. When all the blood samples are collected a laboratory technician and a biochemist will determine the levels of the above mentioned substances, these data will then undergo statistical evaluation.

ELIGIBILITY:
Inclusion Criteria:

* All patients affected by primary inguinal hernia

Exclusion Criteria:

* Diabetes
* Corticosteroids treatment
* Immunosuppressive drugs
* Cirrhotic patients
* Chronic inflammatory disease
* Neoplastic patients

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients affected by primary inguinal hernia
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2010-03; Primary Completion 2010-09 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
Immune response assessment | 0, 6h, 72h and 12 days
  Cytokine measurements

SECONDARY OUTCOMES:
Oxidative stress evaluation | 0, 6h, 24h, 48h and 12 days
  GSH, lipid hydroperoxides and isoprostanes levels

CONTACTS AND LOCATIONS:
Overall Officials: Marcello Donati, MD, PhD, Principal Investigator — University of Catania; Angelo Donati, MD, Study Director — University of Catania
Locations (1):
- University Hospital of Catania, Catania, Italy

REFERENCES:
- [Background] 1) Agarwal BB, et al. Prospective double-blind randomized controlled study comparing heavy- and lightweight polypropylene mesh in totally extraperitoneal repair of inguinal hernia: early results.Surg Endosc. 2009 Feb;23(2):242-7. Epub 2008 Oct 16. 2) Di Vita G, et al. Impact of different texture of polypropylene mesh on the inflammatory response. Int J Immunopathol Pharmacol. 2008 Jan-Mar;21(1):207-14. 3) Cobb WS, Burns JM, et. al. Textile analysis of heavy weight, mid-weight, and light weight polypropylene mesh in a porcine ventral hernia model.J Surg Res. 2006 Nov;136(1):1-7. Epub 2006 Sep 22. 4) Weyhe D, Schmitz I, et al. Experimental comparison of monofile light and heavy polypropylene meshes: less weight does not mean less biological response. World J Surg. 2006 Aug;30(8):1586-91. 5) Di Vita G, Balistreri CR, et al. Systemic inflammatory response in erderly patients following hernioplastical operation. Immun Ageing. 2006 Mar 29;3:3. 6) Di Vita G, Patti R, et al. Acute phase response in oldest-old individuals after surgical stress. J Am Geriatr Soc. 2006 Mar;54(3):561-3. 7) Di Vita G, D'Agostino P, et al. Acute inflammatory response after inguinal and incisional hernia repair with implantation of polypropylene mesh of different size. Langenbecks Arch Surg. 2005 Aug;390(4):306-11. Epub 2005 Feb 3. 8) Brancato G, Gandolfo L, et al. [Biologic tolerance of prolene prosthesis in inguinal hernia repair] Chir Ital. 2003 Sep-Oct;55(5):707-13. 9) Di Vita G, Milano S,et al. Cytokine modifications after tension-free hernioplasty or open conventional inguinal hernia repair. Am J Surg. 2001 Jun;181(6):487-91. 10) Di Vita G, Milano S, et al. Tension-free hernia repair is associated with an increase in inflammatory response markers against the mesh. Am J Surg. 2000 Sep;180(3):203-7. 11) Gürleyik E, Gürleyik G, et al. The inflammatory response to open tension-free inguinal hernioplasty versus conventional repairs. Am J Surg. 1998 Mar;175(3):179-82.
- [Derived] Donati M, Brancato G, Grosso G, Li Volti G, La Camera G, Cardi F, Basile F, Donati A. Immunological reaction and oxidative stress after light or heavy polypropylene mesh implantation in inguinal hernioplasty: A CONSORT-prospective, randomized, clinical trial. Medicine (Baltimore). 2016 Jun;95(24):e3791. doi: 10.1097/MD.0000000000003791. PMID 27310955